CLINICAL TRIAL: NCT06638047
Title: Early Clinical and Radiological Outcomes of a Novel Robotic TKA System
Acronym: RA-TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Tian Hua, MD, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JUST-RA-TKA
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Total Knee Anthroplasty; Robotic Surgery
Keywords: total knee arthroplasty; robot; radiological; clinical outcome; postoperative alignment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RA TKA (Experimental): Robotic-assisted TKA
  Interventions: Procedure: robotic-assisted TKA
- CI TKA (Active Comparator): TKA with conventional instruments
  Interventions: Procedure: CI-TKA

INTERVENTIONS:
Procedure: robotic-assisted TKA — Robotic-assisted TKA means that TKA surgery is operated with the guidance of robotic system.
  Arms: RA TKA
Procedure: CI-TKA — TKA operated with conventional instruments
  Arms: CI TKA

SUMMARY:
This study aimed to evaluate the early clinical and radiological outcomes of robot assisted total knee arthroplasty, and to determine the efficiency and safety of its bone resection and implant positioning of the novel robot system.

144 patients undergoing primary TKA were enrolled in this prospective, multicenter RCT conducted in 3 hospitals. The primary outcome was the rate of patients whose postoperative alignment was less than 3° deviated from the planned evaluated by full-length weight-bearing X-rays of the lower limb at 12 weeks postoperatively. Secondary outcomes will include coronal and sagittal alignment of the components, operation times, blood loss, 12-week range of motion(ROM), 12-week postoperative functional outcomes and satisfaction evaluated by the American Knee Society Score (KSS) and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years (including 18 and 85), regardless of gender;
* Patients scheduled for unilateral primary total knee arthroplasty based on the clinical judgment of the study physician;
* The subject or their guardian has been informed of the study, agrees to all terms of the trial, signs an informed consent form approved by the ethics committee, and agrees to participate in the trial.

Exclusion Criteria:

* The side scheduled for surgery has significant hip joint disease, such as substantial bone defects or severe limitations in joint mobility;
* Patients with active infections around the knee joint or systemic infections;
* Discontinuity or severe functional loss of the knee extensor mechanism, painless knee joint fusion, Charcot joint, poor surgical tolerance, or other conditions that may adversely affect surgical prognosis;
* Patients with contraindications for traditional TKA surgery;
* Pregnant or breastfeeding women;
* Patients known to have excessive alcohol consumption or substance abuse; Body mass index (BMI) > 35 kg/m²;
* Patients who have participated in other clinical trials within one month prior to signing the informed consent form;
* Patients with mental or intellectual disabilities that may affect clinical outcome evaluations;
* Patients deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
HKA outliers | 12 weeks post-surgery
  the proportion of patients with a deviation of ≤ 3° between the mechanical axis (hip-knee-ankle angle, or HKA angle) measured from a full-length, frontal-view lower limb X-ray

SECONDARY OUTCOMES:
FFC angle | 12 weeks post-surgery
  frontal femoral component (FFC) angle
outliers of FFC angle | 12 weeks post-surgery
  outliers of frontal femoral component (FFC) angle (>3 degree)
FTC angle | 12 weeks post-surgery
  frontal tibia component (FTC) angle
outliers of FTC angle | 12 weeks post-surgery
  outliers of frontal tibia component (FTC) angle (>3 degree)
LFC angle | 12 weeks post-surgery
  lateral femoral component (LFC) angle
outliers of LFC angle | 12 weeks post-surgery
  outliers of lateral femoral component (LFC) angle (>3 degree)
LTC angle | 12 weeks post-surgery
  lateral tibia component (LTC) angle
outliers of LTC angle | 12 weeks post-surgery
  outliers of lateral tibia component (LTC) angle (>3 degree)
Surgical duration | During operation
  In this study, surgical duration is defined as the time from the first incision to the completion of skin closure
Blood loss | 3 days after surgery
  Postoperative blood loss is calculated using the Gross formula in this study. The Gross equation was used to calculate the total blood loss (mL) as preoperative blood volume×(preoperative HCT level-postoperative HCT level).
ROM | 12 weeks post-surgery
  ROM refers to the maximum passive range of knee motion
Knee Society Score (KSS) | screening and 12 weeks post-surgery.
  The KSS, developed by the American Knee Society, evaluates objective knee indicators, symptoms, patient satisfaction, patient expectations, and functional activities. A total score above 85 is considered excellent, 70-84 is good, 60-69 is fair, and below 60 is poor.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | screening and 12 weeks post-surgery.
  The WOMAC measures knee function in terms of pain, stiffness, and physical function across 25 items. Pain is assessed with five items, stiffness with two items, and physical function with 18 items. Each item is scored from 0 to 4, with higher scores indicating more severe symptoms.
Incidence of adverse events and serious adverse events | Through study completion, an average of 12 weeks
  Throughout the study, any adverse events that occurred were recorded, and the corresponding incidence was calculated.
  Similarly, any serious adverse events that occurred during the study were recorded, and the corresponding incidence was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No